CLINICAL TRIAL: NCT05317065
Title: The Effect of Mindfulness-Based Stress Reduction Program (MBSR) on Stress, Anxiety and Prenatal Attachment in Risky Pregnants
Brief Title: The Effect of Mindfulness-Based Stress Reduction Program (MBSR) in Risky Pregnants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Emine Akca, Clinical Researcher of the Amasya University Midwifery Department, Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Amasya Univesity
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Stress; Pregnancy, High Risk
Keywords: prenatal attachment; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfullness Based Stress Reduction (Experimental): Mindfullness Based Stress Reduction (MBSR) therapy
  Interventions: Behavioral: Mindfullness Based Stress Reduction (MBSR) intervention
- Control (No Intervention): Control

INTERVENTIONS:
Behavioral: Mindfullness Based Stress Reduction (MBSR) intervention — Mindfullness Based Stress Reduction (MBSR) intervention: Monitoring stress and anxiety levels with mindfulness program
  Arms: Mindfullness Based Stress Reduction

SUMMARY:
Risky pregnant women need various physical and mental health needs, they need to be informed and supported by health personnel. Mindfulness is a non-judgmental and accepting focus of one's attention on what is happening right now. A total of 100 pregnant women (50 experimental, 50 control) are planned to be included in the study. Data will be collected with "Descriptive Information Form", "Prenatal Distress Scale (PBL)-Revised Version", "Pregnancy-Related Anxiety Scale-Revision 2" and "Prenatal Attachment Inventory". In the study, a stress reduction program (MBSR) based on mindfulness will be applied by the researcher to the pregnant women in the experimental group.

DETAILED DESCRIPTION:
Risky pregnancies are a situation that can negatively affect the health of the mother and the fetus, result in the loss of the baby, and bring about physical, social and mental changes. Mindfulness-based approaches have been used in solving both physical and mental problems in pregnant women and very positive results have been obtained. The aim of this study, which was carried out to determine the effect of mindfulness-based stress reduction program (MBSR) on stress, anxiety and prenatal attachment in high-risk pregnant women, is aimed at creating appropriate intervention programs for high-risk pregnancies and contributing to the improvement of pregnancy outcomes. A total of 100 pregnant women (50 experimental, 50 control) are planned to be included in the study. Data will be collected with "Descriptive Information Form", "Prenatal Distress Scale (PBL)-Revised Version", "Pregnancy-Related Anxiety Scale-Revision 2" and "Prenatal Attachment Inventory". In the study, a stress reduction program (MBSR) based on mindfulness will be applied by the researcher to the pregnant women in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

risky pregnant women

Exclusion Criteria:

mental disabilities

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Pregnant
Enrollment: 94 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Prenatal Distress Scale | At the end of the 1 months
  The minimum score that can be obtained from the scale is "0", the maximum score is "34", and as the score obtained from the scale increases, prenatal distress levels also increase.
Pregnancy-Related Anxiety Scale | At the end of the 1 months
  For primiparas, a minimum of 11 points and a maximum of 55 points is obtained, and for multipars, a minimum of 10 and a maximum of 50 points are obtained. As the score obtained from the scale increases, it is accepted that the level of anxiety in pregnancy is higher.

SECONDARY OUTCOMES:
The Prenatal Attachment Inventory | At the end of the 1 months
  A minimum of 21 and a maximum of 84 points can be obtained from the scale. The increase in the score obtained by the pregnant indicates that the level of attachment also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No